CLINICAL TRIAL: NCT03715062
Title: Reducing Antibiotic Prescriptions for Urinary Tract Infection in Long-Term Care Facilities With a Complex Intervention Targeted at Nursing Home Staff -A Protocol for a Cluster Randomized Controlled Trial.
Brief Title: Reducing Antibiotic Prescriptions for Urinary Tract Infection in Long-Term Care Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Unit Of General Practice, Copenhagen (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government); Velux Fonden (Other); Herlev Hospital (Other)
Responsible Party: Principal Investigator, Sif Helene Arnold, Medical Doctor, Research Unit Of General Practice, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 111
Record Dates: First submitted 2018-10-05; First posted 2018-10-22 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Urinary Tract Infections
Keywords: Long-term care facility; ISBAR; Communication; Antibiotics; Antibiotic stewardship
MeSH Terms: conditions — Urinary Tract Infections; Communication | interventions — Observation

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled study, where each Long-term care facility is one cluster.
Masking Description: Statistical analysis is masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receives education in diagnosing urinary tract infection and use of observation, reflection and communication tool.
  Interventions: Other: Dialogue tool
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Dialogue tool — The intervention has two parts: an educational session and a dialogue tool. The educational session consists of 75 minutes of education in diagnosing urinary tract infection. The dialogue tool consists of 1) a checking box for the most important symptoms and observations for urinary tract infection 2) an algorithm to evaluate if urinary tract infection is likely based on the present symptoms and observations 3) a list of reflection points to evaluate with a collegue 4) a specialized ISBAR (communication tool) if long-term care facility staff finds it appropriate to contact the General Practicioner
  Other Names: Observation, reflection and communication tool
  Arms: Intervention group

SUMMARY:
This cluster randomized controlled study evaluates the effect of a tailored observation, reflection and communication tool on used by long-term care facility staff on antibiotic prescription for urinary tract infection in long-term care facility residents.

DETAILED DESCRIPTION:
Healthcare-associated infections due to antimicrobial use in long-term care facilities (LTCF) is an increasing problem in europe. It is well established that there exists a positive correlation between the amount of antibiotics used in treatment and resistant bacteria in both individual patients and society as a whole. A point-prevalence audit from 2017 in LTCFs showed that 10.5% of all LTCF residents in Denmark are treated with an antibiotic agent. In 78% of the cases, the cause for treatment was urinary tract infection (UTI). In addition, this group of elderly are particularly vulnerable to healthcare-associated infections, drug interactions and adverse effects. Thus, there are persuasive reasons for reducing antibiotic use in this specific group.

In the diagnostic process for UTI in a LTCF resident, there are several non-clinical factors influencing the diagnosis and leading to unnecessary treatment. First, because of dementia, sequelae from apoplexies, difficulties walking and other ailments, the typical LTCF resident is unable to express symptoms clearly and attend the GPs office. Consequently, the diagnosis is based on observations made by LTCF staff, which are then communicated to the General Practitioner (GP). Second, the prevalence of asymptomatic bacteriuria is up to 50% in this particular group. Though several studies have found that asymptomatic bacteriuria is a benign condition, it continues to be treated. Third, unspecific symptoms such as mental status change, falls or decreased function are unlikely to be caused by UTI. However, unspecific symptoms are still driving diagnosis and treatment of UTI. These factors may influence diagnosis and treatment in the Danish LTCF setting and therefore, a significant portion of the prescribed antibiotics for UTI could be due to overtreatment.

There is some evidence suggesting that antibiotic stewardship programs focusing on education of LTCF staff decreases antibiotic prescriptions and increases adherence to guidelines. In addition, there is moderate evidence that the widely used communication tool ISBAR (Identification, Situation, Background, Analysis, Recommendation) improves patient safety by improving interprofessional communication especially when communicating over the phone. Thus, if LTCF staff were educated on relevant observation, how to approach ASB, unspecific symptoms and structured handover of clinical information, the impact of these factors on diagnosis and treatment of UTI in LTCF residents may decrease. Overall, antibiotic stewardship programs in LTCF are somewhat effective. However, most of these were targeted at prescribers only or prescribers and nurses and some were also prone to bias because of the choice of study design. At present, there exists no cluster Randomized Controlled Trials (cRCT) targeting only LTCF staff with nursing tasks through a combined education- and communication-centered intervention.

ELIGIBILITY:
Inclusion Criteria:

* LTCFs eligible for inclusion have common service areas with attending staff 24 hours a day and they cannot be specialized i.e. not psychiatric LTCFs or LTCFs for the blind, except for LTCFs specialized in dementia. The residents living in these types of facilities requires a level of care that typically ensures that the LTCF staff handles all contact with the GP on behalf of the resident, while the LTCF residents remains a somewhat homogenous group.
* We include only social and health helpers, social and health assistants and nurses, who have a permanent contract at the LTCF and do day- or evening shifts for the educational session. It is optional for the LTCF to use the educational material to educate LTCF staff in nightshifts. However, a UTI is rarely observed and reported during the night, which is why we chose this pragmatic approach. Usually, if a UTI is suspected, the night shift will report to the day shift, who then reevaluates and contacts the GP if necessary. We also target the permanently employed, as they are the majority of employees with nursing responsibilities and set the standard for the temporary staff.
* All incidents of suspected UTI in LTCF residents or antibiotic prescriptions for UTI must be registered. All registrations must be made on LTCF residents above 65 years of age and with a permanent address at the LTCF, otherwise the incidence of ASB is different than assumed in preparing the intervention.

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1491 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Prescription of antibiotics for urinary tract infection | 17 weeks
  The number of antibiotic prescriptions for urinary tract infections pr resident days

SECONDARY OUTCOMES:
Hospitalization | 17 weeks
  The number of hospitalizations caused by urinary tract infections pr resident days
Death | 17 weeks
  The number of deaths caused by urinary tract infections pr resident days
Appropriate prescription of antibiotics for urinary tract infections | 17 weeks
  The number of treatments with adequate symptoms and observations for treatment pr resident days

OTHER OUTCOMES:
Symptoms | 17 weeks
  The number of symptoms observed in each arm
Observations | 17 weeks
  The number of observations observed in each arm
Contact to doctor | 17 weeks
  Number of times the doctor was contacted pr resident

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bjerrum, MD, PHD, Study Chair — Professor
Locations (1):
- Research Unit of General Practice, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arnold SH, Nygaard Jensen J, Bjerrum L, Siersma V, Winther Bang C, Brostrom Kousgaard M, Holm A. Effectiveness of a tailored intervention to reduce antibiotics for urinary tract infections in nursing home residents: a cluster, randomised controlled trial. Lancet Infect Dis. 2021 Nov;21(11):1549-1556. doi: 10.1016/S1473-3099(21)00001-3. Epub 2021 Jul 22. PMID 34303417
- [Derived] Arnold SH, Jensen JN, Kousgaard MB, Siersma V, Bjerrum L, Holm A. Reducing Antibiotic Prescriptions for Urinary Tract Infection in Nursing Homes Using a Complex Tailored Intervention Targeting Nursing Home Staff: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2020 May 8;9(5):e17710. doi: 10.2196/17710. PMID 32383679